CLINICAL TRIAL: NCT03402633
Title: Leucotrichia in Vitiligo Patients : A Cross Sectional Study
Brief Title: Leucotrichia in Vitiligo
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha Fathy Elmasry, principal investigator, Cairo University
Other Study IDs: Dermatology5
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Leucotrichia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Examination of leukotrichia in vitiligo patients — Examination of leukotrichia will be enhanced by wood's light and dermoscopy for better enhancing of the lesions and good magnification

SUMMARY:
The incidence of leucotrichia has been reported to range from 9 to 48.4% of all vitiligo patients.Leucotrichia is more often observed in segmental vitiligo with a very high percentage. However, further studies considering the prevalence of leucotrichia in different types of vitiligo need to be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Vitiligo patients with/ without leukotrichia within the vitiliginous areas

Exclusion criteria:

* Age < 18
* Premature hair graying in the trunk before the age of 30

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Vitiligo patients with/ without leukotrichia within the vitiliginous areas presenting to dermatology outpatient clinic at Kasr Alainy Teaching Hospital
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Detection of prevalence of leukotrichia within vitilignous areas in vitiligo patients | within 6 months
  Detection of prevalence of leukotrichia within vitilignous areas in vitiligo patients